CLINICAL TRIAL: NCT00164450
Title: TBTC Study 26 PK: Rifapentine Pharmacokinetics in Children Receiving Once Weekly Rifapentine and Isoniazid for the Treatment of Latent Tuberculosis Infection
Brief Title: TBTC Study 26 PK: Rifapentine Pharmacokinetics in Children During Treatment of Latent TB Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: William R. Mac Kenzie, MD, Medical Officer, Tuberculosis Trials Consortiu, DTBE, CDC
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCHSTP-4679
Record Dates: First submitted 2005-09-10; First posted 2005-09-14 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Tuberculosis
Keywords: tuberculosis; TB; pharmacokinetics; children
MeSH Terms: conditions — Tuberculosis | interventions — rifapentine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rifapentine + isoniazid once weekly for 3 months

SUMMARY:
Compared to adults, children appear to require higher weight-based doses of rifapentine to acheive comparable drug levels. TBTC Study 26, a study of the effectiveness and tolerability of weekly rifapentine/isoniazid for three months versus daily isoniazid for nine months for the treatment of latent tuberculosis infection, has been amended to include children ages 2-11 based on an initial single-dose study and pharmacokinetic modeling. Study 26PK evaluates the adequacy of the doses chosen for young children enrolled in Study 26 with a single blood draw, 24 hours after the third or subsequent weekly Study 26 dose of rifapentine and isoniazid. An adult control is enrolled for each child enrolled.

DETAILED DESCRIPTION:
The pharmacokinetics of rifapentine have been studied in adults, adolescents (ages 12-15 years), and patients with hepatic dysfunction and HIV infection. However, there are no published data on the efficacy, safety or pharmacokinetics of rifapentine in children. This lack of data has precluded till now enrollment of children less than 12 years old in TBTC Study 26, a study of the effectiveness and tolerability of weekly rifapentine/isoniazid for three months versus daily isoniazid for nine months for the treatment of latent tuberculosis infection, a phase 3 treatment trial that will enroll 8000 persons with latent tuberculosis infection. A recently completed initial evaluation of rifapentine pharmacokinetics among children receiving a single dose of rifapentine demonstrated significantly lower exposures of rifapentine among children compared to adults, when children were given weight-based doses chosen to be comparable to a 600 mg oral dose in adults. This reduced exposure suggested that children require higher weight-based doses than adults and a model was constructed to estimate rifapentine doses in children that would result in exposures similar to the 900 mg dose used for adults in Study 26. Study 26 has been amended to include children ages 2-11 based on the initial single-dose study and pharmacokinetic modeling. The purpose of Study 26PK is to evaluate the adequacy of the doses chosen for young children who enrolled in Study 26.

Briefly, this study aims to:

* determine whether rifapentine exposure is equivalent in young children receiving weight-based dosing to adults receiving 900 mg.
* correlate rifapentine exposure with toxicity in young children
* validate accuracy of weight-based dosing in children
* determine rifapentine bioavailability in children
* determine association in adults between polymorphisms of MDR1 genotype and rifapentine exposure
* correlate isoniazid concentrations in adults with acetylator status

ELIGIBILITY:
Inclusion Criteria:

1. Enrolled in TBTC Study 26 randomized to treatment with once weekly isoniazid and rifapentine:

   * Child between the ages of 2 to less than 12 years for whom informed consent by a guardian and of assent (if applicable) have been obtained.
   * Adult greater than age 18 for whom informed consent has been obtained.
2. Willingness to undergo a blood phlebotomy 24 hours following dosing of isoniazid and rifapentine after receiving at least three once-weekly doses of rifapentine plus isoniazid.

If as a result of a contact investigation, both a parent and child are enrolled in Study 26, both may be co-enrolled into the pharmacokinetic substudy with the adult serving as the control for the child. Preference will be given to a biologic parent of the same gender. If no eligible biologic parent is available for study, the next adult of the same gender and at the same TBTC site, who is substudy eligible, will serve as the adult control.

Exclusion Criteria:

* None

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2005-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Determine whether rifapentine exposure (level 24 hours after drug ingestion) is equivalent in young children receiving weight-based dosing to adults receiving 900 mg. | 24 hours after drug ingestion

SECONDARY OUTCOMES:
Correlate estimated rifapentine exposure with toxicity in young children receiving rifapentine and isoniazid for latent tuberculosis infection. | During the three months of taking rifapentine
Validate the accuracy of estimated rifapentine exposure with pediatric rifapentine dose based on weight. | 24 hours after drug ingestion
Determine estimated drug bioavailability in pediatric subjects (ages 2 to < 12 years) given higher mg/kg doses of rifapentine. | 24 hours after drug ingestion
Determine the association in adults between polymorphisms of MDR1 genotype (P-glycoprotein) and rifapentine estimated exposure. | at the time of blood draw
Determine the frequency of lower antitubercular drug concentrations in adults with acetylator status determined by N-acetyltransferase genotypes and of rifapentine by C24 and by MDR1 genotypes. | at the time of blood draw

CONTACTS AND LOCATIONS:
Overall Officials: Marc Weiner, MD, Study Chair — VAMC and University of Texas Health Science Center San Antonio
Locations (24):
- United States (19):
  - Central Arkansas Veterans Health System, Little Rock, Arkansas
  - University of Southern California Medical Center, Los Angeles, California
  - University of California at San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Denver Public Health Department, Denver, Colorado
  - Washington DC Veterans Administration Medical Center, Washington D.C., District of Columbia
  - Emory University School of Medicine, Atlanta, Georgia
  - Northwestern University School of Medicine, Chicago, Illinois
  - Hines Veterans Administration Medical Center, Hines, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston University Medical Center, Boston, Massachusetts
  - New Jersey School of Medicine, Newark, New Jersey
  - Columbia University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Veterans Administration Tennessee Valley Health Care System, Nashville, Tennessee
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Houston Veterans Administration Medical Center, Houston, Texas
  - Audie L. Murphy VA Hospital, San Antonio, Texas
  - Seattle-King County Health Department, Seattle, Washington
- Hopital Universitario Clementino Fraga Filho, Rio de Janeiro, Rio de Janeiro, Brazil
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnepeg, Manitoba
  - Montreal Chest Institute, Montreal, Quebec
- Agencia de Salut Publica, Barcelona, Spain